CLINICAL TRIAL: NCT02623725
Title: Immunogenicity and Safety of a Tetravalent Dengue Vaccine Given as a Booster Injection in Adolescents and Adults Who Previously Completed the 3-dose Schedule in a Study Conducted in Latin America
Brief Title: Study of a Booster Dose of a Tetravalent Dengue Vaccine in Subjects Who Previously Completed the 3-dose Schedule
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CYD64; U1111-1161-2855 (Other: WHO)
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever
Keywords: Dengue Fever; Dengue virus; Dengue Hemorrhagic Fever; CYD Dengue Vaccine
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Dosage Forms; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An observer-blind procedure was followed for the injection of the CYD Dengue Vaccine booster or placebo. Neither the observer Investigator, nor the Sponsor, nor the participant/participants' parent(s)/legally acceptable representative(s) knew which product was administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CYD Dengue Vaccine Booster Group (Experimental): Participants who received 3 doses of the tetravalent dengue vaccine in previous CYD dengue vaccine studies (CYD13 or CYD30), received a booster injection of CYD dengue vaccine at Day 0 in this study (CYD64).
  Interventions: Biological: CYD Dengue Vaccine (5-dose formulation)
- Placebo Group (Experimental): Participants who received 3 doses of the tetravalent dengue vaccine in previous CYD dengue vaccine studies (CYD13 or CYD30), received an injection of placebo at Day 0 in this study (CYD64).
  Interventions: Biological: Placebo, NaCl 0.9%

INTERVENTIONS:
Biological: CYD Dengue Vaccine (5-dose formulation) — 0.5 mL, Subcutaneous
  Arms: CYD Dengue Vaccine Booster Group
Biological: Placebo, NaCl 0.9% — 0.5 mL, Subcutaneous
  Arms: Placebo Group

SUMMARY:
The aim of the study was to assess and describe the booster effect of a CYD dengue vaccine dose administered 4 to 5 years after the completion of a 3-dose vaccination schedule.

Primary Objective

- To demonstrate the non-inferiority, in terms of geometric mean of titer ratios (GMTRs), of a CYD dengue vaccine booster compared to the third CYD dengue vaccine injection in participants from CYD13 - NCT00993447 and CYD30 - NCT01187433 trials (participants from Group 1 only).

Secondary Objectives:

* If the primary objective of non-inferiority was achieved: To demonstrate the superiority, in terms of GMTRs, of a CYD dengue vaccine booster compared to the third CYD dengue vaccine injection in participants from CYD13 and CYD30 trials.
* To describe the immune responses elicited by a CYD dengue vaccine booster and placebo injection in participants who received 3 doses of the CYD dengue vaccine in the CYD13 and CYD30 trials in all participants.
* To describe the neutralizing antibody levels of each dengue serotype post-dose 3 (CYD13 and CYD30 participants) and immediately prior to booster or placebo injection in all participants.
* To describe the neutralizing antibody persistence 6 months, 1 year, and 2 years post booster or placebo injection in all participants.
* To evaluate the safety of booster vaccination with the CYD dengue vaccine in all participants.

DETAILED DESCRIPTION:
Healthy adolescents and adults who received 3 doses of the tetravalent dengue vaccine 4 to 5 years earlier in previous CYD dengue vaccine trials (CYD13 and CYD30) received either a booster dose CYD dengue vaccine or a placebo on Day 0. They were evaluated for safety and antibody persistence of the booster injection up to 2 years post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Had been identified as a potential participant by the Sponsor and is included in the list provided to the Investigator (i.e., aged 9 to 16 years on the day of first vaccination of CYD dengue vaccine in CYD13/CYD30 and has a post-dose 3 serum sample available [at least 400 microliters of serum]).
* Participants were in good health, based on medical history and physical examination.
* Assent form or informed consent form (ICF) had been signed and dated by the participant (based on local regulations), and ICF had been signed and dated by the parent(s) or another legally acceptable representative (and by an independent witness if required by local regulations).
* Participant and parent(s)/legally acceptable representative(s) attended all scheduled visits and complied with all trial procedures.

Exclusion Criteria:

* Participant who received any other dengue vaccination that was not part of the CYD13 or CYD30 trials.
* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination).
* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following the trial vaccination.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with trial conduct or completion.
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature >= 38.0°C). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 251 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2018-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (5):
- Investigational Site Number 001, Vitória, Brazil
- Investigational Site Number 002, Bucaramanga, Colombia
- Investigational Site Number 003, Tegucigalpa, Honduras
- Investigational Site Number 004, Temixco, Mexico
- Investigational Site Number 005, Carolina, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Coronel D, Garcia-Rivera EJ, Rivera M, Arredondo-Garcia JL, Dietze R, Perroud AP, Cortes M, Bonaparte M, Zhao J, Tila M, Jackson N, Zambrano B, Noriega F. Dengue Vaccine Booster in Healthy Adolescents and Adults in Latin America: Evaluation 4-5 Years After a Primary 3-Dose Schedule. Pediatr Infect Dis J. 2019 May;38(5):e90-e95. doi: 10.1097/INF.0000000000002286. PMID 30986790
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 14 April 2016 to 19 October 2016 at 5 sites, one each in Brazil, Colombia, Honduras, Mexico, and Puerto Rico.
Pre-assignment Details: A total of 251 participants who received 3 doses of CYD dengue vaccine in previous studies CYD13 (NCT00993447) and CYD30 (NCT01187433) were enrolled and randomized in this study (CYD64).
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Started | 187 | 64
Completed | 171 | 58
Not Completed | 16 | 6
Not completed — Non compliance with protocol | 9 | 3
Not completed — Serious adverse event | 0 | 2
Not completed — Withdrawal by Subject | 7 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group | Total
Number analyzed (Participants) | 187 | 64 | 251
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 63 | 19 | 82
  Between 18 and 65 years | 124 | 45 | 169
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.2 (2.14) | 19.0 (1.99) | 19.1 (2.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 27 | 116
  Male | 98 | 37 | 135

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers of Antibodies Against Each Dengue Virus Serotype Following Booster Injection With CYD Dengue Vaccine in CYD64 Compared to Third CYD Dengue Vaccine Received in CYD13/CYD30: CYD Dengue Vaccine Booster Group
Description: Geometric Mean Titers (GMTs) of antibodies against each of the 4 dengue virus serotype (parental strains) were assessed using the plaque reduction neutralization test (PRNT).
Time Frame: 28 days post-dose 3 in CYD13 or CYD30 and 28 days post-booster injection in CYD64
Population: Analysis was performed on Per-Protocol Analysis Set which included all participants who had no protocol deviations from the present study (CYD64). Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Groups:
- CYD Dengue Vaccine Booster Group:Post Dose 3 in CYD13 or CYD30: Participants who received 3 doses of the tetravalent dengue vaccine in previous CYD dengue vaccine studies (CYD13 or CYD30) were included in this study (CYD64).
- CYD Dengue Vaccine Booster Group: Post Booster Dose in CYD64: Participants who received 3 doses of the tetravalent dengue vaccine in previous CYD dengue vaccine studies (CYD13 or CYD30), received a booster injection of CYD dengue vaccine at Day 0 in this study (CYD64).
Arm/Group | CYD Dengue Vaccine Booster Group:Post Dose 3 in CYD13 or CYD30 | CYD Dengue Vaccine Booster Group: Post Booster Dose in CYD64
Number analyzed (Participants) | 177 | 177
titers (1/dilution)
  Dengue Virus Serotype 1: number analyzed (Participants) | 176 | 177
  Dengue Virus Serotype 1 | 316 [233 to 428] | 560 [421 to 744]
  Dengue Virus Serotype 2: number analyzed (Participants) | 175 | 177
  Dengue Virus Serotype 2 | 356 [275 to 462] | 657 [520 to 830]
  Dengue Virus Serotype 3: number analyzed (Participants) | 175 | 177
  Dengue Virus Serotype 3 | 640 [516 to 794] | 671 [535 to 843]
  Dengue Virus Serotype 4: number analyzed (Participants) | 176 | 177
  Dengue Virus Serotype 4 | 243 [195 to 303] | 344 [279 to 424]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Booster Group:Post Dose 3 in CYD13 or CYD30 vs CYD Dengue Vaccine Booster Group: Post Booster Dose in CYD64; Dengue Virus Serotype 1; Test type: Non-Inferiority — The overall non-inferiority of the booster dose was to be demonstrated if the lower limit of the two-sided 95 percent (%) Confidence Interval (CI) of the Geometric mean of titer ratios (GMTRs) (booster vs post-dose 3) was greater than (>) 1/2 for each serotype; Geometric mean of titer ratio = 1.66, 95% CI 2-sided [1.33 to 2.06]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Booster Group:Post Dose 3 in CYD13 or CYD30 vs CYD Dengue Vaccine Booster Group: Post Booster Dose in CYD64; Dengue Virus Serotype 2; Test type: Non-Inferiority — The overall non-inferiority of the booster dose was to be demonstrated if the lower limit of the two-sided 95% CI of the GMTRs (booster vs post-dose 3) was >1/2 for each serotype; Geometric mean of titer ratio = 1.82, 95% CI 2-sided [1.43 to 2.31]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine Booster Group:Post Dose 3 in CYD13 or CYD30 vs CYD Dengue Vaccine Booster Group: Post Booster Dose in CYD64; Dengue Virus Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Geometric mean of titer ratio = 1.04, 95% CI 2-sided [0.841 to 1.27]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine Booster Group:Post Dose 3 in CYD13 or CYD30 vs CYD Dengue Vaccine Booster Group: Post Booster Dose in CYD64; Dengue Virus Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Geometric mean of titer ratio = 1.32, 95% CI 2-sided [1.01 to 1.74]

2. Secondary Outcome: GMTs of Antibodies Against Each Dengue Virus Serotype Following Booster Injection With CYD Dengue Vaccine in CYD64 Compared to Third CYD Dengue Vaccine Received in CYD13/CYD30: CYD Dengue Vaccine Booster Group
Description: GMTs of antibodies against each of the 4 dengue virus serotype (parental strains) following booster injection were assessed using PRNT.
Time Frame: 28 days post-dose 3 in CYD13 or CYD30 and 28 days post-booster injection in CYD64
Population: Analysis was performed on Full analysis set which included all participants who received either CYD Dengue Vaccine or placebo and had blood sample drawn and valid post-injection serology results. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Booster Group:Post Dose 3 in CYD13 or CYD30 | CYD Dengue Vaccine Booster Group: Post Booster Dose in CYD64
Number analyzed (Participants) | 184 | 184
titers (1/dilution)
  Dengue Virus Serotype 1: number analyzed (Participants) | 183 | 184
  Dengue Virus Serotype 1 | 304 [225 to 409] | 538 [406 to 714]
  Dengue Virus Serotype 2: number analyzed (Participants) | 182 | 184
  Dengue Virus Serotype 2 | 338 [261 to 436] | 648 [515 to 817]
  Dengue Virus Serotype 3: number analyzed (Participants) | 182 | 184
  Dengue Virus Serotype 3 | 617 [499 to 762] | 660 [528 to 827]
  Dengue Virus Serotype 4: number analyzed (Participants) | 183 | 184
  Dengue Virus Serotype 4 | 241 [195 to 298] | 341 [278 to 418]
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Booster Group:Post Dose 3 in CYD13 or CYD30 vs CYD Dengue Vaccine Booster Group: Post Booster Dose in CYD64; Dengue Virus Serotype 1; Test type: Superiority — The superiority was to be demonstrated if the lower limit of the two-sided 95% CI for the ratio was >1; Geometric mean of titer ratio = 1.66, 95% CI 2-sided [1.34 to 2.05]
Statistical Analysis 2: Comparison: CYD Dengue Vaccine Booster Group:Post Dose 3 in CYD13 or CYD30 vs CYD Dengue Vaccine Booster Group: Post Booster Dose in CYD64; Dengue Virus Serotype 2; Test type: Superiority — The superiority was to be demonstrated if the lower limit of the two-sided 95% CI for the ratio was >1; Geometric mean of titer ratio = 1.89, 95% CI 2-sided [1.49 to 2.41]
Statistical Analysis 3: Comparison: CYD Dengue Vaccine Booster Group:Post Dose 3 in CYD13 or CYD30 vs CYD Dengue Vaccine Booster Group: Post Booster Dose in CYD64; Dengue Virus Serotype 3; Test type: Superiority — The superiority was to be demonstrated if the lower limit of the two-sided 95% CI for the ratio was >1; Geometric mean of titer ratio = 1.06, 95% CI 2-sided [0.860 to 1.30]
Statistical Analysis 4: Comparison: CYD Dengue Vaccine Booster Group:Post Dose 3 in CYD13 or CYD30 vs CYD Dengue Vaccine Booster Group: Post Booster Dose in CYD64; Dengue Virus Serotype 4; Test type: Superiority — The superiority was to be demonstrated if the lower limit of the two-sided 95% CI for the ratio was >1; Geometric mean of titer ratio = 1.33, 95% CI 2-sided [1.02 to 1.73]

3. Secondary Outcome: GMTs of Antibodies Against Each Dengue Virus Serotype Before And Following Booster Injection (Inj.) With Either CYD Dengue Vaccine or Placebo
Description: as for outcome 2
Time Frame: Pre-booster injection (Day 0) and 28 days post-booster injection
Population: Analysis was performed on Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 177 | 64
titers (1/dilution)
  Dengue Virus Serotype 1: Pre-booster Inj. | 325 [233 to 452] | 349 [201 to 607]
  Dengue Virus Serotype 1: 28 days Post-booster Inj. | 560 [421 to 744] | 297 [162 to 547]
  Dengue Virus Serotype 2: Pre-booster Inj. | 360 [267 to 484] | 323 [195 to 535]
  Dengue Virus Serotype 2: 28 days Post-booster Inj. | 657 [520 to 830] | 354 [205 to 610]
  Dengue Virus Serotype 3: Pre-booster Inj. | 357 [269 to 472] | 442 [270 to 724]
  Dengue Virus Serotype 3: 28 days Post-booster Inj. | 671 [535 to 843] | 432 [266 to 700]
  Dengue Virus Serotype 4: Pre-booster Inj. | 162 [134 to 195] | 161 [108 to 242]
  Dengue Virus Serotype 4: 28 days Post-booster Inj. | 344 [279 to 424] | 161 [110 to 237]

4. Secondary Outcome: GMTRs of Antibodies Against Each Dengue Virus Serotype Before and Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: GMTs of antibodies against each of the 4 dengue virus serotype (parental strains) following booster injection were assessed using PRNT. GMTRs were calculated as the ratio of GMTs post-booster injection and pre-booster injection.
Time Frame: Pre-booster injection (Day 0) and 28 days post-booster injection
Population: Analysis was performed on Per-Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 177 | 64
ratio
  Dengue Virus Serotype 1 | 1.59 [1.33 to 1.90] | 0.798 [0.623 to 1.02]
  Dengue Virus Serotype 2 | 1.70 [1.43 to 2.03] | 1.03 [0.754 to 1.40]
  Dengue Virus Serotype 3 | 1.78 [1.47 to 2.16] | 0.946 [0.749 to 1.19]
  Dengue Virus Serotype 4 | 2.09 [1.65 to 2.63] | 0.946 [0.777 to 1.15]

5. Secondary Outcome: Percentage of Participants With Seropositivity Against Each Dengue Virus Serotype Before and Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: Seropositivity against each dengue virus serotype were measured using dengue PRNT. Seropositive participants were defined as the participants with neutralizing antibody titers greater than or equal to (>=)10 (1/dilution).
Time Frame: Pre-booster injection (Day 0) and 28 days post-booster injection
Population: Analysis was performed on Per-Protocol Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 177 | 64
percentage of participants
  Dengue Virus Serotype 1: Pre-booster Inj. | 88.1 | 90.6
  Dengue Virus Serotype 1: 28 days Post-booster Inj. | 96.0 | 84.4
  Dengue Virus Serotype 2: Pre-booster Inj. | 89.8 | 90.6
  Dengue Virus Serotype 2: 28 days Post-booster Inj. | 98.9 | 87.5
  Dengue Virus Serotype 3: Pre-booster Inj. | 92.1 | 95.3
  Dengue Virus Serotype 3: 28 days Post-booster Inj. | 99.4 | 95.3
  Dengue Virus Serotype 4: Pre-booster Inj. | 97.2 | 92.2
  Dengue Virus Serotype 4: 28 days Post-booster Inj. | 100.0 | 93.8

6. Secondary Outcome: Percentage of Participants With Seroconversion Against Each Dengue Virus Serotype Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: Seroconversion for each serotype was defined as the percentage of participants with either a pre-booster titer <10 (1/dilution) and a post-booster titer >=40 (1/dilution), or a pre-booster titer >=10 (1/dilution) and a >=4-fold increase in post-booster titer as determined by PRNT.
Time Frame: 28 days post-booster injection
Population: Analysis was performed on Full analysis set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 184 | 64
percentage of participants
  Dengue Virus Serotype 1 | 17.9 | 3.1
  Dengue Virus Serotype 2 | 20.1 | 17.2
  Dengue Virus Serotype 3 | 21.2 | 4.7
  Dengue Virus Serotype 4 | 20.7 | 6.3

7. Secondary Outcome: GMTs of Antibodies Against Each Dengue Virus Serotype Following the Third CYD Dengue Vaccine Injection Received in Study CYD13/CYD30, and Before Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: GMTs of antibodies against each of the 4 dengue virus serotype (parental strains) were assessed using the PRNT.
Time Frame: 28 days post-dose 3 in CYD13 or CYD30 and pre-booster injection (Day 0) in CYD64
Population: Analysis was performed on Per-Protocol Analysis Set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 177 | 64
titers (1/dilution)
  Dengue Virus Serotype 1: 28 days Post-dose 3: number analyzed (Participants) | 176 | 64
  Dengue Virus Serotype 1: 28 days Post-dose 3 | 316 [233 to 428] | 232 [142 to 381]
  Dengue Virus Serotype 1: Pre-booster Inj. | 325 [233 to 452] | 349 [201 to 607]
  Dengue Virus Serotype 2: 28 days Post-dose 3: number analyzed (Participants) | 175 | 64
  Dengue Virus Serotype 2: 28 days Post-dose 3 | 356 [275 to 462] | 303 [210 to 438]
  Dengue Virus Serotype 2: Pre-booster Inj. | 360 [267 to 484] | 323 [195 to 535]
  Dengue Virus Serotype 3: 28 days Post-dose 3: number analyzed (Participants) | 175 | 64
  Dengue Virus Serotype 3: 28 days Post-dose 3 | 640 [516 to 794] | 541 [372 to 785]
  Dengue Virus Serotype 3: Pre-booster Inj. | 357 [269 to 472] | 442 [270 to 724]
  Dengue Virus Serotype 4: 28 days Post-dose 3: number analyzed (Participants) | 176 | 63
  Dengue Virus Serotype 4: 28 days Post-dose 3 | 243 [195 to 303] | 255 [192 to 340]
  Dengue Virus Serotype 4: Pre-booster Inj. | 162 [134 to 195] | 161 [108 to 242]

8. Secondary Outcome: GMTRs of Antibodies Against Each Dengue Virus Serotype Following the Third CYD Dengue Vaccine Injection Received in Study CYD13/CYD30, and Before Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: GMTs of antibodies against each of the 4 dengue virus serotype (parental strains) were assessed using the PRNT. GMTRs were calculated as the ratio of GMTs pre-booster injection and post-dose injection.
Time Frame: 28 days post-dose 3 in CYD13 or CYD30 and pre-booster injection (Day 0) in CYD64
Population: Analysis was performed on Per-Protocol Analysis Set. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 177 | 64
ratio
  Dengue Virus Serotype 1: number analyzed (Participants) | 176 | 64
  Dengue Virus Serotype 1 | 0.952 [0.765 to 1.18] | 1.41 [0.927 to 2.14]
  Dengue Virus Serotype 2: number analyzed (Participants) | 175 | 64
  Dengue Virus Serotype 2 | 0.986 [0.778 to 1.25] | 1.04 [0.662 to 1.65]
  Dengue Virus Serotype 3: number analyzed (Participants) | 175 | 64
  Dengue Virus Serotype 3 | 0.536 [0.440 to 0.654] | 0.818 [0.574 to 1.16]
  Dengue Virus Serotype 4: number analyzed (Participants) | 176 | 63
  Dengue Virus Serotype 4 | 0.618 [0.497 to 0.770] | 0.613 [0.427 to 0.881]

9. Secondary Outcome: Percentage of Participants With Seropositivity Against Each Dengue Virus Serotype Following the Third CYD Dengue Vaccine Injection Received in Study CYD13/CYD30, and Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: Seropositivity against each dengue virus serotype were measured using dengue PRNT. Seropositive participants were defined as the participants with neutralizing antibody titers >=10 (1/dilution).
Time Frame: 28 days post-dose 3 in CYD13 or CYD30 and 28 days post-booster injection in CYD64
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 177 | 64
percentage of participants
  Dengue Virus Serotype 1: 28 days Post-dose 3: number analyzed (Participants) | 176 | 64
  Dengue Virus Serotype 1: 28 days Post-dose 3 | 90.9 | 90.6
  Dengue Virus Serotype 1: 28 days Post-booster Inj. | 96.0 | 84.4
  Dengue Virus Serotype 2: 28 days Post-dose 3: number analyzed (Participants) | 175 | 64
  Dengue Virus Serotype 2: 28 days Post-dose 3 | 95.4 | 96.9
  Dengue Virus Serotype 2: 28 days Post-booster Inj. | 98.9 | 87.5
  Dengue Virus Serotype 3: 28 days Post-dose 3: number analyzed (Participants) | 175 | 64
  Dengue Virus Serotype 3: 28 days Post-dose 3 | 100.0 | 100.0
  Dengue Virus Serotype 3: 28 days Post-booster Inj. | 99.4 | 95.3
  Dengue Virus Serotype 4: 28 days Post-dose 3: number analyzed (Participants) | 176 | 63
  Dengue Virus Serotype 4: 28 days Post-dose 3 | 92.0 | 96.8
  Dengue Virus Serotype 4: 28 days Post-booster Inj. | 100.0 | 93.8

10. Secondary Outcome: GMTs of Antibodies Against Each Dengue Virus Serotype Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: as for outcome 2
Time Frame: 6 months,12 months, and 24 months post-booster injection in CYD64
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 177 | 64
titers (1/dilution)
  Dengue Virus Serotype 1:6 months Post-booster Inj.: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 1:6 months Post-booster Inj. | 270 [205 to 356] | 192 [111 to 329]
  Dengue Virus Serotype1:12 months Post-booster Inj.: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype1:12 months Post-booster Inj. | 270 [205 to 356] | 185 [112 to 304]
  Dengue Virus Serotype1:24 months Post-booster Inj.: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype1:24 months Post-booster Inj. | 241 [180 to 323] | 182 [112 to 297]
  Dengue Virus Serotype 2:6 months Post-booster Inj.: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 2:6 months Post-booster Inj. | 442 [358 to 546] | 335 [217 to 515]
  Dengue Virus Serotype2:12 months Post-booster Inj.: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype2:12 months Post-booster Inj. | 269 [217 to 335] | 225 [152 to 334]
  Dengue Virus Serotype2:24 months Post-booster Inj.: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype2:24 months Post-booster Inj. | 246 [192 to 315] | 187 [126 to 279]
  Dengue Virus Serotype 3:6 months Post-booster Inj.: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 3:6 months Post-booster Inj. | 503 [397 to 636] | 447 [285 to 701]
  Dengue Virus Serotype3:12 months Post-booster Inj.: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype3:12 months Post-booster Inj. | 303 [242 to 379] | 328 [219 to 491]
  Dengue Virus Serotype3:24 months Post-booster Inj.: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype3:24 months Post-booster Inj. | 341 [275 to 423] | 309 [194 to 492]
  Dengue Virus Serotype 4:6 months Post-booster Inj.: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 4:6 months Post-booster Inj. | 233 [198 to 273] | 156 [115 to 212]
  Dengue Virus Serotype4:12 months Post-booster Inj.: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype4:12 months Post-booster Inj. | 169 [144 to 199] | 127 [96.3 to 167]
  Dengue Virus Serotype4:24 months Post-booster Inj.: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype4:24 months Post-booster Inj. | 150 [129 to 174] | 114 [85.2 to 153]

11. Secondary Outcome: GMTRs of Antibodies Against Each Dengue Virus Serotype Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: as for outcome 4
Time Frame: Pre-booster injection (Day 0), 6 months, 12 months, and 24 months post-booster injection in CYD64
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 177 | 64
ratio
  Dengue Virus Serotype 1: Month 6/Day 0: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 1: Month 6/Day 0 | 0.763 [0.643 to 0.904] | 0.502 [0.364 to 0.693]
  Dengue Virus Serotype 1: Month 12/Day 0: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype 1: Month 12/Day 0 | 0.722 [0.607 to 0.859] | 0.483 [0.366 to 0.638]
  Dengue Virus Serotype 1: Month 24/Day 0: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype 1: Month 24/Day 0 | 0.642 [0.532 to 0.774] | 0.509 [0.382 to 0.678]
  Dengue Virus Serotype 2: Month 6/Day 0: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 2: Month 6/Day 0 | 1.14 [0.922 to 1.40] | 0.998 [0.716 to 1.39]
  Dengue Virus Serotype 2: Month 12/Day 0: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype 2: Month 12/Day 0 | 0.651 [0.539 to 0.786] | 0.630 [0.460 to 0.863]
  Dengue Virus Serotype 2: Month 24/Day 0: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype 2: Month 24/Day 0 | 0.579 [0.473 to 0.709] | 0.548 [0.373 to 0.806]
  Dengue Virus Serotype 3: Month 6/Day 0: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 3: Month 6/Day 0 | 1.34 [1.09 to 1.65] | 0.957 [0.701 to 1.31]
  Dengue Virus Serotype 3: Month 12/Day 0: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype 3: Month 12/Day 0 | 0.786 [0.652 to 0.947] | 0.667 [0.505 to 0.883]
  Dengue Virus Serotype 3: Month 24/Day 0: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype 3: Month 24/Day 0 | 0.878 [0.749 to 1.03] | 0.682 [0.523 to 0.890]
  Dengue Virus Serotype 4: Month 6/Day 0: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 4: Month 6/Day 0 | 1.42 [1.17 to 1.72] | 0.912 [0.691 to 1.20]
  Dengue Virus Serotype 4: Month 12/Day 0: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype 4: Month 12/Day 0 | 1.02 [0.846 to 1.22] | 0.709 [0.553 to 0.909]
  Dengue Virus Serotype 4: Month 24/Day 0: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype 4: Month 24/Day 0 | 0.890 [0.753 to 1.05] | 0.684 [0.534 to 0.877]

12. Secondary Outcome: Percentage of Participants With Seropositivity Against Each Dengue Virus Serotype Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: as for outcome 9
Time Frame: 6 months,12 months, and 24 months post-booster injection in CYD64
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 177 | 64
percentage of participants
  Dengue Virus Serotype 1:6 months Post-booster Inj.: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 1:6 months Post-booster Inj. | 91.4 | 85.7
  Dengue Virus Serotype1:12 months Post-booster Inj.: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype1:12 months Post-booster Inj. | 92.9 | 88.7
  Dengue Virus Serotype1:24 months Post-booster Inj.: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype1:24 months Post-booster Inj. | 87.2 | 89.7
  Dengue Virus Serotype 2:6 months Post-booster Inj.: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 2:6 months Post-booster Inj. | 98.9 | 92.1
  Dengue Virus Serotype2:12 months Post-booster Inj.: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype2:12 months Post-booster Inj. | 96.5 | 91.9
  Dengue Virus Serotype2:24 months Post-booster Inj.: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype2:24 months Post-booster Inj. | 93.3 | 91.4
  Dengue Virus Serotype 3:6 months Post-booster Inj.: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 3:6 months Post-booster Inj. | 97.7 | 95.2
  Dengue Virus Serotype3:12 months Post-booster Inj.: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype3:12 months Post-booster Inj. | 97.1 | 96.8
  Dengue Virus Serotype3:24 months Post-booster Inj.: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype3:24 months Post-booster Inj. | 99.4 | 94.8
  Dengue Virus Serotype 4:6 months Post-booster Inj.: number analyzed (Participants) | 174 | 63
  Dengue Virus Serotype 4:6 months Post-booster Inj. | 98.9 | 95.2
  Dengue Virus Serotype4:12 months Post-booster Inj.: number analyzed (Participants) | 170 | 62
  Dengue Virus Serotype4:12 months Post-booster Inj. | 97.6 | 95.2
  Dengue Virus Serotype4:24 months Post-booster Inj.: number analyzed (Participants) | 164 | 58
  Dengue Virus Serotype4:24 months Post-booster Inj. | 98.8 | 94.8

13. Secondary Outcome: Number of Participants Reporting Solicited Injection Site Reactions (Pain, Erythema, Swelling) Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Grade 3 reactions: Pain: significant; prevents daily activity; Erythema and Swelling: >100 millimeters (mm).
Time Frame: Within 7 days after booster injection
Population: Analysis was performed on Safety Analysis Set which included all participants who received either CYD dengue vaccine or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 187 | 64
Participants
  Injection-site Pain: Any | 46 | 12
  Injection-site Pain: Grade 3 | 1 | 0
  Injection-site Erythema: Any | 1 | 0
  Injection-site Erythema: Grade 3 | 0 | 0
  Injection-site Swelling: Any | 0 | 0
  Injection-site Swelling: Grade 3 | 0 | 0

14. Secondary Outcome: Number of Participants Reporting Solicited Systemic Reactions (Fever, Headache, Malaise, Myalgia, Asthenia) Following Booster Injection With Either CYD Dengue Vaccine or Placebo
Description: Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Grade 3 reactions: Fever: >=39°C; Headache, Malaise, Myalgia, and Asthenia: significant, prevents daily activity.
Time Frame: Within 14 days after booster injection
Population: Analysis was performed on Safety Analysis Set. Here, 'number analyzed' = participants with available data for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
Number analyzed (Participants) | 187 | 64
Participants
  Fever: Any Grade: number analyzed (Participants) | 179 | 63
  Fever: Any Grade | 13 | 6
  Fever: Grade 3: number analyzed (Participants) | 179 | 63
  Fever: Grade 3 | 1 | 1
  Headache: Any Grade | 87 | 22
  Headache: Grade 3 | 11 | 2
  Malaise: Any Grade | 47 | 19
  Malaise: Grade 3 | 5 | 0
  Myalgia: Any Grade | 60 | 19
  Myalgia: Grade 3 | 2 | 2
  Asthenia: Any Grade | 52 | 14
  Asthenia: Grade 3 | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected from Day 0 (post-vaccination) up to 28 days post-booster injection. Solicited Reaction (SR) data was collected within 7 and 14 days after vaccination. Serious adverse event (SAE) data was collected throughout the study (up to 24 months after last vaccination).
Description: Analysis was performed on Safety Analysis Set. A SR was an AE that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination.
Arm/Group | CYD Dengue Vaccine Booster Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/187 | 2/64
Serious Adverse Events (participants affected / at risk) | 19/187 | 5/64
Other Adverse Events (participants affected / at risk) | 115/187 | 31/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Booster Group (N=187) | Placebo Group (N=64)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Abortion Induced (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Booster Group (N=187) | Placebo Group (N=64)
Asthenia (General disorders) | 52 (52) | 14 (14)
Injection Site Pain (General disorders) | 46 (46) | 12 (12)
Malaise (General disorders) | 47 (48) | 19 (19)
Pyrexia (General disorders) | 15 (15) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 60 (61) | 19 (19)
Headache (Nervous system disorders) | 88 (90) | 22 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.